CLINICAL TRIAL: NCT06270251
Title: Modeling Tic Change During Behavior Therapy for Tics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSYCH-2023-32292
Record Dates: First submitted 2024-01-30; First posted 2024-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Tic Disorder
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Youth ages 12-21 years with chronic tics will complete a course of 10 outpatient, weekly CBIT sessions with pre-, post-, 1-month and 3-month follow up assessments.
  Interventions: Behavioral: CBIT

INTERVENTIONS:
Behavioral: CBIT — 8sessions of CBIT following a published treatment manual delivered over 10 weeks (the last two sessions are biweekly)
  CBIT is a well-established behavioral treatment that is considered by the American Academy of Neurology to be the first-line intervention for tics.

SUMMARY:
Chronic tics are a disabling neuropsychiatric symptom associated with multiple child-onset mental disorders. Chronic tics affect 1-3% of youth and can be associated with impaired functioning, emotional and behavioral problems, physical pain, diminished quality of life, and peer victimization. Chronic tics are the primary symptom of Tourette Syndrome (TS) and Persistent Motor/Vocal Tic Disorders.

CBIT is a manualized treatment focused on increasing tic controllability. Its core procedure is competing response training (CRT), in which patients learn to inhibit tics by learning and applying a competing motor action to one tic at a time. CBIT is recommended as a first-line treatment relative to medications and other therapies. However, only 52% of children and 38% of adults show clinically meaningful tic improvement. Large randomized trials have demonstrated the superiority of CBIT over supportive therapy in child and adult patients, and meta-analysis shows comparable effect sizes for CBIT and medication. Although increasing tic controllability is the primary goal of CBIT, tic controllability nor its correlates have been examined longitudinally during the intervention.

The overall objective of this study is to use fine-grained data collection strategies to identify patterns in tic controllability and other relevant related variables that are associated with treatment response to CBIT. Participants with chronic tics will complete a manualized course of 8-session CBIT. Behavioral, psychosocial, and global functioning will be assessed longitudinally to examine predictors and correlates of response. CBIT sessions will be video recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-21 years at time of enrollment.
* Current chronic motor and/or vocal tics, defined as tics for at least 1 year without a tic-free period of more than 3 consecutive months. Tics must not be due to a medical condition or the direct physiological effects of a substance.
* At least moderate tic severity, defined as a Yale Global Tic Severity Scale total score

  ≥14 (≥9 for those with motor or vocal tics only).
* Full scale IQ greater than 70
* English fluency to ensure comprehension of study measures and instructions.

Exclusion Criteria:

* Active suicidality.
* Previous diagnosis of psychosis or cognitive disability.
* Substance abuse or dependence within the past year.
* Concurrent psychotherapy focused on tics.
* Neuroleptic/antipsychotic medications.
* Taking a medication that has not reached stability criterion (same medication and dose for 6 weeks with no planned changes over the intervention period)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Tic Severity | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Yale Global Tic Severity Scale (YGTSS) will be used, which is Gold-standard, clinician administered tic severity scale. It includes symptom checklist of specific tic types YGTSS ranges from 0-50, higher scores are more severe tic symptoms
Sheehan Disability scale | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Self and parent measure of functional impairment
Behavior Rating Inventory of Executive Function | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Self and parent-rated measure of impairment of executive function
Ask Suicide-Screening Questions (ASQ) | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Clinician-administered screen of suicidality
Child Attitudes Toward Illness Scale (CATIS) | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Self-report measure of favorably or unfavorably adolescent feels about having a chronic illness
Rosenberg Self-Esteem Scale | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Self-report measure of adolescent feelings of self-esteem and self-worth
Caregiver Strain Questionnaire | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Measure of strain experienced by caregivers and family of youth with health/emotional challenges
Clinical Global Impressions (CGI) | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Clinician, patient, parent-rated global measure of illness severity and improvement
Parent/Adult Tic Questionnaire | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Adult-self or parent-report measure of tic symptoms and severity

SECONDARY OUTCOMES:
Premonitory Urge for Tics Scale | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Self-report measure of intensity of urges to tic
Tic Suppression Task | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Direct observation measure of tic suppression ability
Stop signal task | Baseline, post-treatment (week 8-10), follow up 1 (week 4-6 post-treatment) and follow up 2 (week 12-14) post-treatment)
  Computerized task measuring ability to inhibit prepotent motor responses. This task is optional.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Conelea, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States